CLINICAL TRIAL: NCT04191317
Title: Pain Neuroscience Education and Gradual Exposure to Exercise in Factory Workers With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Doctor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-CED/2019
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Two arms, each receiving a different intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education and gradual exposure (Experimental): Education explaining the neurophysiological processes that lead to chronic pain, in order to change maladaptive belief towards disease, reconceptualising them and desensitizing the Central Nervous system.
  On first session of gradual exposure the patients are challenged to create a hierarchically list with the functional activities they experience fear, and exposure begins with the one they have less. Both the therapist and participant will determine a specific group of exercises after the patient understands the benign nature of pain, and will be evaluated the maximal performance of the individual to perform each exercise separately.
  Interventions: Other: Pain Neuroscience Education and gradual exposure
- Pilates and postural education (Active Comparator): In the first session, basic Pilates principles will be taught and reinforced at the beginning of the follow up sessions, including: postural alignment (neutral spine position, shoulder blade and neck position) and core recruitment along with a controlled breathing. Each session will have a warm up, mobility, stability and strengthening exercises and a cool down period.
  Interventions: Other: Pilates and postural education

INTERVENTIONS:
Other: Pain Neuroscience Education and gradual exposure — Education covering the pathophysiology of apin and exercises based on the gradual exposure principle
  Arms: Pain Neuroscience Education and gradual exposure
Other: Pilates and postural education — Postural education and pilates exercises
  Arms: Pilates and postural education

SUMMARY:
This study aims to compare the effectiveness of a pain neuroscience education (PNE) based programe and gradual exposure to exercise versus pilates on disability levels associated with chronic low back pain in factory workers. There will be two arms each one receiving one type of intervention over 8 weeks.

DETAILED DESCRIPTION:
This will be a pilot randomized controlled and experimental study. There will be two groups, one group will receive an intervention strategy based in basic postural re-education exercises (Pilates) and self-management strategies, and the other group will perform a program based in pain neuroscience education and gradual exposure to exercise. Both interventions will be delivered in the physiotherapy office of a paper industry. Participants will be randomly allocated according to the work team they belong, to an intervention arm.

The inclusion criteria to participate in the study are: to have nonspecific low back pain lasting longer than three months, felt in the anatomic region below the costal margin and above the inferior gluteal folds, without referred leg pain and not related to any specific pathology such as lumbar fracture, ankylosing spondylitis, cauda equina syndrome, infection or tumour and not receiving treatment for low back pain. Participants will be excluded if during the physical examination they show altered sensorial signs indicative of radiculopathy; red flags such as weight loss without a particular cause, cancer diagnosis or sustained use of corticoids; presence of any rheumatic, neurologic or cardiorespiratory disease that prevent the practice of physical exercise.

Once inclusion criteria have been ascertained, participants will be assessed for sociodemographic and anthropometric data, pain, disability, knowledge of pain neurophysiology, pain catastrophizing, fear of movement, presence of a neuropathic component, workstation evaluation and global impression of change related to intervention.

The intervention will last for 8 weeks, during which participants will have 1 face-to-face session per week with a duration of approximately 60 minutes each. One group (Pilates group) will receive an intervention based on Pilates' and and postural education. The other group will have theoretical sessions of PNE and gradual exposure to exercise (PNE plus graded exposure group).

ELIGIBILITY:
Inclusion Criteria:

* to have nonspecific low back pain lasting longer than three months, felt in the anatomic region below the costal margin and above the inferior gluteal folds, without referred leg pain and not related to any specific pathology such as lumbar fracture, ankylosing spondylitis, cauda equina syndrome, infection or tumour;
* not receiving treatment for low back pain.

Exclusion Criteria:

* altered sensorial signs indicative of radiculopathy; red flags such as weight loss without a particular cause, cancer diagnosis or sustained use of corticoids;
* presence of any rheumatic, neurologic or cardiorespiratory disease that prevent the practice of physical exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline (week 0)
  Measured using the Numerical Rating Scale (NRS), a 11-point scale is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst pain imaginable)
Pain intensity | End of study - week 9
  Measured using the Numerical Rating Scale (NRS), a 11-point scale is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst pain imaginable)
Pain intensity | 3 months follow up
  Measured using the Numerical Rating Scale (NRS), a 11-point scale is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Disability | Baseline (week 0)
  Measured using the Roland Morris Disability Questionnaire, scored a minimum of 0 and a maximum of 24
Disability | End of study - week 9
  Measured using the Roland Morris Disability Questionnaire, scored a minimum of 0 and a maximum of 24
Disability | 3 months follow up
  Measured using the Roland Morris Disability Questionnaire, scored a minimum of 0 and a maximum of 24
Knowledge of pain neurophysiology | Baseline - week 0
  Measured using the Neurophysiology of Pain Questionnaire scored a minimum of 0 and a maximum of 19
Knowledge of pain neurophysiology | End of study - week 9
  Measured using the Neurophysiology of Pain Questionnaire scored a minimum of 0 and a maximum of 19
Knowledge of pain neurophysiology | 3 months follow up
  Measured using the Neurophysiology of Pain Questionnaire scored a minimum of 0 and a maximum of 19
Pain catastrophizing | Baseline - week 0
  Measured using the Pain Catastrophizing Scale scored a minimum of 0 and a maximum of 52
Pain catastrophizing | End of study - week 9
  Measured using the Pain Catastrophizing Scale scored a minimum of 0 and a maximum of 52
Pain catastrophizing | 3 months follow up
  Measured using the Pain Catastrophizing Scale scored a minimum of 0 and a maximum of 52
Fear avoidance behavior | Baseline - week 0
  Measured using the Tampa Scale of Kinesiophobia, total score varies from 13 to 52, where 13 represents the less and 52 the greater level of fear of movement
Fear avoidance behavior | End of study - week 9
  Measured using the Tampa Scale of Kinesiophobia, total score varies from 13 to 52, where 13 represents the less and 52 the greater level of fear of movement
Fear avoidance behavior | 3 months follow up
  Measured using the Tampa Scale of Kinesiophobia, total score varies from 13 to 52, where 13 represents the less and 52 the greater level of fear of movement
Pain phenotype | Baseline - week 0
  Measured using the Pain Detect Questionnaire. Total score varies from -1 to 38 points. Scores below 12 indicate little probability of a neuropathic component (85% chance of not having); scores between 12 - 19 reveal a mixed phenotype, whereas a score above 19 reveals high probability of neuropathic pain (90% chance).
Pain phenotype | End of study - week 9
  Measured using the Pain Detect Questionnaire. Total score varies from -1 to 38 points. Scores below 12 indicate little probability of a neuropathic component (85% chance of not having); scores between 12 - 19 reveal a mixed phenotype, whereas a score above 19 reveals high probability of neuropathic pain (90% chance).
Pain phenotype | 3 months follow up
  Measured using the Pain Detect Questionnaire. Total score varies from -1 to 38 points. Scores below 12 indicate little probability of a neuropathic component (85% chance of not having); scores between 12 - 19 reveal a mixed phenotype, whereas a score above 19 reveals high probability of neuropathic pain (90% chance).
Patient Global Impression of Change | Baseline - week 0
  Measured using the Patient Global Impression of Change (PGIC) scale. This is a unidimensional measure widely used in chronic pain studies, in which the patients classify their improvements using a 7-point scale, varying from "1- no change" to "7 - a great deal better and a considerable improvement that has made all the difference"
Patient Global Impression of Change | End of study - week 9
  Measured using the Patient Global Impression of Change (PGIC) scale. This is a unidimensional measure widely used in chronic pain studies, in which the patients classify their improvements using a 7-point scale, varying from "1- no change" to "7 - a great deal better and a considerable improvement that has made all the difference"
Patient Global Impression of Change | 3 months follow up
  Measured using the Patient Global Impression of Change (PGIC) scale. This is a unidimensional measure widely used in chronic pain studies, in which the patients classify their improvements using a 7-point scale, varying from "1- no change" to "7 - a great deal better and a considerable improvement that has made all the difference"

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No